CLINICAL TRIAL: NCT04126317
Title: A Randomized, Single-Masked, Active-Controlled Phase 2 Study of the Safety, Tolerability, and Efficacy of Repeated Doses of High-Dose Aflibercept in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Safety, Tolerability, and Efficacy of Aflibercept in Patients With Neovascular Age-Related Macular Degeneration
Acronym: CANDELA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGFTe (HD)-AMD-1905
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Neovascular (Wet) Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-masked: The patients, visual acuity examiners, imaging technicians and reading center will be masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- intravitreal aflibercept injection (IAI) (Experimental): Treatment-naïve patients with neovascular "wet" age-related macular degeneration (nAMD) randomized in a 1:1 ratio
  Interventions: Drug: aflibercept
- High-dose aflibercept (HD) (Experimental): Treatment-naïve patients with nAMD randomized in a 1:1 ratio
  Interventions: Drug: High-dose aflibercept

INTERVENTIONS:
Drug: aflibercept — Intravitreally (IVT) administered as a liquid formulation in a vial
  Other Names: EYLEA®; BAY86-5321
  Arms: intravitreal aflibercept injection (IAI)
Drug: High-dose aflibercept — Intravitreally (IVT) administered as a liquid formulation in a vial
  Arms: High-dose aflibercept (HD)

SUMMARY:
The primary objectives of the study are to determine the safety of high-dose aflibercept (hereafter referred to as HD) and to determine if HD provides greater intraocular pharmacodynamic (PD) effect and/or longer duration of action compared to intravitreal aflibercept injection (hereafter referred to as IAI).

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women ≥50 years of age with active subfoveal choroidal neovascularization (CNV) secondary to nAMD
* Best Corrected Visual Acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score of 78 to 24 (Snellen equivalent of 20/32 to 20/320) in the study eye

Key Exclusion Criteria:

* Evidence of CNV due to any cause other than nAMD in either eye
* Evidence of diabetic macular edema (DME) or diabetic retinopathy (defined as more than 1 microaneurysm) in either eye in diabetic patients
* Prior use of IVT anti-VEGF agents (aflibercept, ranibizumab, bevacizumab, brolucizumab, pegaptanib sodium) in the study eye
* Prior IVT investigational agents in either eye (eg, anti-ang-2/anti-VEGF bispecific monoclonal antibodies, gene therapy)
* Previous use of intraocular or periocular corticosteroids within 120 days of screening or treatment with an IVT steroid implant at any time in the study eye
* History of vitreoretinal surgery (including scleral buckling) in the study eye
* Any other intraocular surgery within 12 weeks (84 days) before the screening visit
* History of corneal transplant or corneal dystrophy in study eye

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (46):
- United States (45):
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Sun City, Arizona
  - Regeneron Study Site, Encino, California
  - Regeneron Study Site, Fullerton, California
  - Regeneron Study Site, Mountain View, California
  - Regeneron Study Site, Palm Desert, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, Santa Ana, California
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Golden, Colorado
  - Regeneron Study Site, Waterford, Connecticut
  - Regeneron Study Site, Fort Lauderdale, Florida
  - Regeneron Study Site, Fort Myers, Florida
  - Regeneron Study Site, Lakeland, Florida
  - Regeneron Study Site, Largo, Florida
  - Regeneron Study Site, Melbourne, Florida
  - Regeneron Study Site, Tallahassee, Florida
  - Regeneron Study Site, Winter Haven, Florida
  - Regeneron Study Site, Augusta, Georgia
  - Regeneron Study Site, Marietta, Georgia
  - Regeneron Study Site, Oak Forest, Illinois
  - Regeneron Study Site, Hagerstown, Maryland
  - Regeneron Study Site, Royal Oak, Michigan
  - Regeneron Study Site, Bloomfield, New Jersey
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, Albuquerque, New Mexico
  - Regeneron Study Site, Great Neck, New York
  - Regeneron Study Site, Asheville, North Carolina
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Edmond, Oklahoma
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Kingston, Pennsylvania
  - Regeneron Study Site, Ladson, South Carolina
  - Regeneron Study Site, West Columbia, South Carolina
  - Regeneron Study Site, Rapid City, South Dakota
  - Regeneron Study Site, Abilene, Texas
  - Regeneron Study Site, Arlington, Texas
  - Regeneron Study Site, Austin, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, The Woodlands, Texas
  - Regeneron Study Site, Salt Lake City, Utah
  - Regeneron Study Site, Fairfax, Virginia
  - Regeneron Study Site, Spokane, Washington
  - Regeneron Study Site, Morgantown, West Virginia
- Regeneron Study Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Wykoff CC, Brown DM, Reed K, Berliner AJ, Gerstenblith AT, Breazna A, Abraham P, Fein JG, Chu KW, Clark WL, Leal S, Schmelter T, Hirshberg B, Yancopoulos GD, Vitti R; CANDELA Study Investigators. Effect of High-Dose Intravitreal Aflibercept, 8 mg, in Patients With Neovascular Age-Related Macular Degeneration: The Phase 2 CANDELA Randomized Clinical Trial. JAMA Ophthalmol. 2023 Sep 1;141(9):834-842. doi: 10.1001/jamaophthalmol.2023.2421. PMID 37535382

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 245 participants screened, 106 participants were randomized and treated.
Groups:
- Intravitreal Aflibercept Injection (IAI): Treatment-naïve participants with neovascular "wet" age-related macular degeneration (nAMD) were randomized in a 1:1 ratio to receive IAI (2 mg) monthly for 3 initial injections (baseline, week 4, and week 8), followed by additional doses at weeks 20 and 32.
- High-Dose Aflibercept Injection (HD): Treatment-naïve participants with nAMD were randomized in a 1:1 ratio to receive HD aflibercept (8 mg) monthly for 3 initial injections (baseline, week 4, and week 8), followed by additional doses at weeks 20 and 32.
Period: Overall Study
Arm/Group | Intravitreal Aflibercept Injection (IAI) | High-Dose Aflibercept Injection (HD)
Started | 53 | 53
Completed | 49 | 51
Not Completed | 4 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravitreal Aflibercept Injection (IAI) | High-Dose Aflibercept Injection (HD) | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (8.27) | 77.0 (7.69) | 77.4 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 30 | 66
  Male | 17 | 23 | 40
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic of Latino | 4 | 2 | 6
    Not Hispanic or Latino | 49 | 51 | 100
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 51 | 52 | 103
    American Indian or Alaska Native | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Other | 1 | 0 | 1
Number of Participants without Retinal Fluid in the Center Subfield of Study Eye [Count of Participants; unit: Participants] — Center subfield=the circular area in 1 millimeter (mm) diameter centered around the center point of the fovea. Without fluid defined as absence of intraretinal fluid (IRF) and/or subretinal fluid (SRF) in the center subfield. Presence of retinal fluid was assessed by spectral domain optical coherence tomography (SD-OCT)
  Participants | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Time Frame: Up to Week 44
Population: Safety analysis set (SAF): All randomized participants who received any study drug; it was based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreal Aflibercept Injection (IAI) | High-Dose Aflibercept Injection (HD)
Number analyzed (Participants) | 53 | 53
Participants
  Participants with at least 1 Ocular TEAE of the Study Eye | 20 | 20
  Participants with at least 1 Ocular TEAE of the Fellow Eye | 13 | 13
  Participants with at least 1 Non-Ocular TEAE | 24 | 28

2. Primary Outcome: Number of Participants With at Least One Serious TEAE
Time Frame: Up to Week 44
Population: SAF: All randomized participants who received any study drug; it was based on the treatment received (as treated)
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreal Aflibercept Injection (IAI) | High-Dose Aflibercept Injection (HD)
Number analyzed (Participants) | 53 | 53
Participants
  Participants with at least 1 Ocular Serious TEAE of the Study Eye | 1 | 2
  Participants with at least 1 Ocular Serious TEAE of the Fellow Eye | 0 | 0
  Participants with at least 1 Non-Ocular Serious TEAE | 4 | 5

3. Primary Outcome: Number of Participants Without Retinal Fluid in the Center Subfield of Study Eye
Description: Center subfield=the circular area in 1 millimeter (mm) diameter centered around the center point of the fovea. Without fluid defined as absence of intraretinal fluid (IRF) and/or subretinal fluid (SRF) in the center subfield. Presence of retinal fluid was assessed by spectral domain optical coherence tomography (SD-OCT)
Time Frame: At Week 16
Population: Full analysis set (FAS): All randomized participants; it was based on the treatment allocated (as randomized). Missing post-baseline values for a given participant were imputed using the last observation carried forward (LOCF).
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreal Aflibercept Injection (IAI) | High-Dose Aflibercept Injection (HD)
Number analyzed (Participants) | 53 | 53
Participants | 18 | 27

ADVERSE EVENTS:
Time Frame: From first dose up to Week 44 (end of study)
Arm/Group | Intravitreal Aflibercept Injection (IAI) | High-Dose Aflibercept Injection (HD)
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/53
Serious Adverse Events (participants affected / at risk) | 4/53 | 7/53
Other Adverse Events (participants affected / at risk) | 14/53 | 19/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Aflibercept Injection (IAI) (N=53) | High-Dose Aflibercept Injection (HD) (N=53)
Chest pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Retinal tear Study Eye (Eye disorders) | 0 (0) | 1 (1)
Visual impairment Study Eye (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced Study Eye (Eye disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Aflibercept Injection (IAI) (N=53) | High-Dose Aflibercept Injection (HD) (N=53)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Conjunctival haemorrhage Fellow Eye (Eye disorders) | 1 (1) | 3 (3)
Neovascular age-related macular degeneration Fellow Eye (Eye disorders) | 3 (3) | 4 (4)
Vitreous detachment Fellow Eye (Eye disorders) | 3 (3) | 1 (2)
Conjunctival haemorrhage Study Eye (Eye disorders) | 2 (2) | 3 (3)
Neovascular age-related macular degeneration Study Eye (Eye disorders) | 4 (4) | 2 (2)
Vitreous detachment Study Eye (Eye disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT04126317/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04126317/SAP_001.pdf